CLINICAL TRIAL: NCT07362173
Title: Actualities in Procedural Sedation: Remimazolam
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Iuliu Hatieganu University of Medicine and Pharmacy (Other)
Collaborators: Institutul Regional de Gastroenterologie & Hepatologie Prof. dr. Octavian Fodor (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 5129/29.04.2025, AVZ213/21.07
Record Dates: First submitted 2025-07-04; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2025-07

CONDITIONS: ASA Class III/IV Patients; COPD III/IV; Age 65 and Older; Multiple Organ Failure
MeSH Terms: conditions — Multiple Organ Failure

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Remimazolam (Active Comparator): Lot 1 - Participants in this arm will receive remimazolam for procedural sedation. Remimazolam will be administered intravenously according to the institutional sedation protocol, with dosing adjusted to achieve adequate procedural sedation.
  Interventions: Drug: Administering remimazolam
- Propofol (Active Comparator): Lot 2 - Participants in this arm will receive Propofol for procedural sedation. Propofol will be administered intravenously according to standard clinical practice, with dosing adjusted to achieve adequate procedural sedation.
  Interventions: Drug: Administering propofol

INTERVENTIONS:
Drug: Administering remimazolam — Administering Remimazolam for procedural sedation
  Arms: Remimazolam
Drug: Administering propofol — Administering Propofol for procedural sedation
  Arms: Propofol

SUMMARY:
Remimazolam is a new, ultra-short-acting benzodiazepine approved in Romania for procedural sedation. It shows significant clinical benefits compared to other sedatives like Propofol or Midazolam, especially in elderly or high-risk patients. Advantages include better hemodynamic stability, reduced respiratory depression, lower incidence of postoperative delirium, and rapid recovery without residual sedation. It is metabolized by liver esterases and is less affected by organ dysfunction. Clinical studies suggest that remimazolam may be a safer and more effective alternative in procedural and general anesthesia. The findings support the development of institutional protocols for its use, particularly in high-risk populations and endoscopic procedures.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 65 years or older
* ASA Physical Status classification III or IV
* Patients scheduled to undergo endoscopic procedures requiring procedural sedation
* Ability to provide written informed consent

Exclusion Criteria:

* Age below 65 years
* Pediatric population
* Refusal or inability to provide informed consent
* Severe allergy to study drugs
* Pregnancy or breastfeeding

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Heart rate (beats per minute) | Periprocedural
  The lowest heart rate will be recorded
Mean arterial pressure (mmHg) | Periprocedural
  The lowest mean arterial pressure will be recorded
Incidence of hypotension requiring vasoactive support (Yes/No) | Periprocedural
  The presence of hypotension requiring vasoactive drug administration will be recorded.

SECONDARY OUTCOMES:
Patient satisfaction | Postprocedural
  Patient satisfaction will be recorded as a single score per participant.
Endoscopist satisfaction (5-point Likert scale) | Periprocedural
  Endoscopist satisfaction will be evaluated and recorded as a single 5-point Likert score per participant.
Quality of recovery (ordinal scale) | Periprocedural
  Quality of recovery will be assessed using an ordinal clinical scale and reported as a single score per participant.
Incidence of postoperative nausea and vomiting (Yes/No) | Periprocedural
  The presence of nausea and/or vomiting will be recorded.
Total dose of sedative administered (mg) | Periprocedural
  Total intravenous dose of the sedative agent administered during the procedure.
Need for airway intervention due to apnea (Yes/No) | Periprocedural
  The need for airway support due to apnea will be recorded.
Incidence of apnea (Yes/No) | Periprocedural
  The occurrence of apnea during procedural sedation will be recorded.
Peripheral oxygen saturation (SpO₂,%) | Periprocedural
  Peripheral capillary oxygen saturation will be measured using pulse oximetry and summarized as the mean periprocedural value.
Respiratory rate (breaths per minute) | Periprocedural
  Respiratory rate will be monitored during the periprocedural period.
Duration of apnea (seconds) | Periprocedural
  Duration of apnea episodes will be measured in seconds.
Need for change in sedation regimen (Yes/No) | Periprocedural
  The need to change the planned sedation regimen will be recorded.
Incidence of postprocedural delirium (Yes/No) | Periprocedural
  Postprocedural delirium or agitation will be recorded.
Incidence of adverse events (Yes/No) | Periprocedural
  The occurrence of adverse events related to procedural sedation will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Regional Institute of Gastroenterology-Hepatology Prof. Dr. Octavian Fodor, Cluj-Napoca, Cluj, Romania

IPD SHARING:
Plan to Share IPD: No
Due to the investigator-initiated nature of the study and local data protection regulations, individual participant data will not be made available for sharing.